CLINICAL TRIAL: NCT01759225
Title: Computerized Registry of Cardiovascular Disease Patients
Brief Title: Registry of Cardiovascular Disease Patients
Acronym: CVD Registry
Status: Enrolling by invitation | Type: Observational
Sponsor: Maccabi Healthcare Services, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: MACCVREG1; cvdregistry (Registry Identifier: Cardiovascular Disease Patients)
Record Dates: First submitted 2012-12-18; First posted 2013-01-03 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Ischemic Heart Disease; Congestive Heart Failure; Peripheral Vascular Disease; Cerebrovascular Disease; Atrial Fibrillation; Cerebrovascular Atherosclerosis
Keywords: Registry, Cardiovascular, CVD, Health Maintenance Organization
MeSH Terms: conditions — Myocardial Ischemia; Heart Failure; Peripheral Vascular Diseases; Cerebrovascular Disorders; Atrial Fibrillation; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month

GROUPS / COHORTS (1):
- Cardiovascular Disease Patients

SUMMARY:
A computerized registry of cardiovascular disease patients in a large health maintenance organization in Israel. The registry is aimed to be used by health professionals to identify cardiovascular disease patients and to follow the courses of their illnesses and risk factors.

DETAILED DESCRIPTION:
The registry was initiated in 1998 by Maccabi Healthcare services, which is the second largest publicly funded HMO in Israel,serving 24% of the total population with a nationwide distribution.

The registry uses advanced information technology that integrates personal computerized community and hospital records, data from laboratory tests, dispensed medications, physiological signals, radiological images, and reports from investigations and procedures.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of the following:

Ischemic Heart Disease,MI,non-MI,congestive heart failure,peripheral vascular disease, cerebrovascular disease CVA,TIA,patients with first AMI diagnosis from community physicians if they were hospitalized for lasting at least 3 days during a 30-day period prior to diagnosis.

* Patients with prior coronary artery bypass grafting(CABG) or percutaneous coronary intervention (PCI), using relevant Current Procedural Terminology (CPT) codes

Exclusion Criteria:

* patients who were diagnosed as suffering from CHD by primary physician or general hospitals prior to 2000 with no further indication
* Patients whose primary physician reported that the patient is CHD-free providing adequate medical records

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The electronic registry includes all patients that had been diagnosed twice or more by hospital or outpatient cardiologists, primary physicians, or pediatricians with at least one of the following clinical diagnoses, classified according to the International Classification of Diseases, Ninth revision (ICD-9) codes: Ischemic Heart Disease,MI,non-MI,congestive heart failure,peripheral vascular disease, cerebrovascular disease CVA,TIA, Patients with prior coronary artery bypass grafting(CABG) or percutaneous coronary intervention (PCI), using relevant Current Procedural Terminology (CPT) codes were also included in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 110000 (Estimated)
Dates: Start 1998-01; Primary Completion 2100-12 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Cardiovascular disease | Up to 100 years

SECONDARY OUTCOMES:
prevalence rates of CVD | up to 100 years
Major Adverse Cardiac Events | up to 100 years
Number of LDL Tests performed reaching target LDL | up to 100 years
Proportion of dyslipidemia patients treated with Statins | up to 100 years

OTHER OUTCOMES:
hospitalization days due to CVD | up to 100 years

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Chodick, PHD, Study Director — Head,Epidemiology & Database Reseaech Unit, Medical Division, Maccabi H.S
Locations (1):
- Maccabi Healthcare Services, Tel Aviv, Israel

REFERENCES:
- [Result] Shalev V, Chodick G, Goren I, Silber H, Kokia E, Heymann AD. The use of an automated patient registry to manage and monitor cardiovascular conditions and related outcomes in a large health organization. Int J Cardiol. 2011 Nov 3;152(3):345-9. doi: 10.1016/j.ijcard.2010.08.002. Epub 2010 Sep 9. PMID 20826019